CLINICAL TRIAL: NCT05212584
Title: CD7 CAR-T Cell Treatment of Relapsed/Refractory CD7+ T -Acute Lymphoblastic Leukemia/ Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: iCell Gene Therapeutics (Industry)
Collaborators: iCar Bio Therapeutics (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ICG170-001
Record Dates: First submitted 2022-01-16; First posted 2022-01-28 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-01

CONDITIONS: Relapsed/Refractory, High Risk Hematologic Malignancies; T-ALL/Lymphoma
Keywords: CD7; CD7CAR; leukemia; acute lymphoblastic leukemia/lymphoma; hematologic malignancies
MeSH Terms: conditions — Recurrence; Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: CD7 CAR T cells are used to treat patients. Patient will be administered either fresh or thawed CAR T cells by IV injection after receiving lymphodepleting chemotherapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD7 CAR T cells (Experimental): Dose escalation phase: CD7 CAR T cells will be transduced with a lentiviral vector to express a CD7 CARs. with an escalation approach, 1 e6 to 7 e6 CAR-T cells/kg
  Interventions: Biological: CD7CAR T cells

INTERVENTIONS:
Biological: CD7CAR T cells — CD7 CAR T cells are used to treat patients. Patient will be administered either fresh or thawed CAR T cells by IV injection after receiving lymphodepleting chemotherapy.

SUMMARY:
This is a phase I, interventional, single arm, open label, treatment study to evaluate the safety and tolerability of CD7 CAR-T cells in patients with relapsed and/or refractory, high risk hematologic malignancies.

DETAILED DESCRIPTION:
T-acute lymphoblast leukemia (T-ALL) accounts for 15-20% of all ALL cases. It is a neoplastic lymphoid leukemia characterized by the proliferation of immature precursor T cells. T-ALL is a highly aggressive tumor. Adults need intensive chemotherapy, and the cure rate is <50%, even with stem cell transplantation. The prognosis is also very poor. The combined chemotherapy has significantly improved the prognosis of T-acute lymphoblast leukemia/lymphoma. However, once the disease appears to be relapsed/refractory, there is limited treatment options, and the overall prognosis is extremely poor. Therefore, exploring safe and effective treatments is a critical unmet medical need. Since 95% of T-ALLs express CD7, this might provide an effective targeting approach for the vast majority of T-ALL cases.

ELIGIBILITY:
Inclusion Criteria:

* 1. Signed written informed consent; Patients volunteer to participate in the clinical trial; 2. Diagnosis is mainly based on the World Health Organization (WHO) 2008; 3. Complete remission cannot be achieved after induction therapy; recurrence occurs after completion remission; the burden of leukemic blasts in the peripheral blood or bone marrow is greater than 5%; 4. Leukemic blast cells express CD7 (CD7 positive by flow cytometry or immunohistochemistry ≥70%); 5. The expected survival period is greater than 12 weeks; 6. ECOG score ≤2; 7. Age 2-60 years old; 8. HGB≥70g/L (can be transfused); 9. Total bilirubin does not exceed 3 times the upper limit of normal value, and AST and ALT do not exceed 5 times the upper limit of normal value.

Exclusion Criteria:

* 1. Patients declining to consent for treatment 2. Prior solid organ transplantation 3. One of the following cardiac issues: atrial fibrillation; myocardial infarction within the past 12 months; prolonged QT syndrome or secondary QT prolongation; clinically significant pericardial effusion; cardiac insufficiency NYHA (New York Heart Association) III or IV; 4. History of severe pulmonary dysfunction diseases; 5. Severe infection or persistent infection cannot be effectively controlled; 6. Severe autoimmune disease or congenital immunodeficiency; 7. Active hepatitis; 8. Human immunodeficiency virus (HIV) infection; 9. Clinically significant viral infections, or uncontrollable viral reactivation, including EBV (Epstein-Barr virus).

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The number and incidence of adverse events after CD7 CAR infusion. | Up to 3 months
  Evaluation all possible adverse reactions, including the number, incidence, and severity of symptoms such as cytokine release syndromes and neurotoxicity within 3 months after CAR infusion

SECONDARY OUTCOMES:
Disease response to CD7 CAR T cells | Up to 1 year
  The disease response to CD7 CAR T cells is evaluated by bone marrow biopsy and aspirate within 1 years after CAR infusion. The proportion of subjects receiving CD7 CAR T infusion to 1) morphological remission (blasts <5%): 2) flow cytometry analysis was blast negative, and 3) molecular biological remission (if applicable).
Evaluation of curative effects | Up to 1 year
  Evaluation of curative effects within 1 year including 1)completion remission (CR), 2) complete remission with incomplete recovery of blood cells (CRi), 3) minimal residual disease positive (MRD+), 4)minimal residual disease negative (MRD-), and 4) disease recurrence or progression
Overall survival | Up to 1 year
  Overall survival {1 year after CAR infusion] . The time from the start of CD7 CAR T injection to death is determined as the overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Peihua Lu, MD, Principal Investigator — Hebei Yanda Lu Daopei Hospital, China
Locations (1):
- Hebei Yanda Lu Daopei Hospital, Langfang, Hebei, China